CLINICAL TRIAL: NCT05614193
Title: Deep Enhanced Imaging in Stroke and Vascular Neurology
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Chairman, Chinese PLA General Hospital
Other Study IDs: AI-301
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Radiology; Cerebral Stroke; Vascular Diseases
Keywords: Deep learning; Medical imaging; Cerebral stroke; Cerebrovascular disease; Vascular imaging
MeSH Terms: conditions — Stroke; Vascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Imaging group: Participants with suspecting brain stroke or vascular lesion conducted conventional CT or MR imaging and deep enhanced imaging.
  Interventions: Diagnostic Test: Deep learning imaging enhancement

INTERVENTIONS:
Diagnostic Test: Deep learning imaging enhancement — Conventional imaging or down-sampling imaging from CT or MR are enhanced by approved deep learning method.

SUMMARY:
To investigate the performance of enhanced computed tomography (CT) or magnetic resonance (MR) imaging by deep learning relative to conventional CT or MR imaging in brain stroke and vascular neurology. We expect that the deep enhanced imaging method can shorten the time stay in the imaging session of stroke patients, optimize the overall imaging quality and improve the patients' care in imaging session.

DETAILED DESCRIPTION:
Early diagnosis of cerebral infarction, detection of ischemic penumbra, evaluation of collateral circulation and identification of vascular lesions by imaging are critical for treatment decision and outcome improvement in cerebral stroke. Multimodal computed tomography (CT) and magnetic resonance (MR) imaging are most prevalent and accessible approaches in clinical scenarios. These two approaches are downgraded either by radiation exposure or long scanning time which may hinder the rapid treatment for patients. Deep learning has shown substantial achievements in medical imaging enhancement. The added value of deep learning method in stroke and vascular neurology has not been thoroughly validated. In this study, we aimed to investigate the performance of enhanced computed tomography (CT) or magnetic resonance (MR) imaging by deep learning relative to conventional CT or MR imaging in brain stroke and vascular neurology. We expect that the deep enhanced imaging method can shorten the time stay in the imaging session of stroke patients, optimize the overall imaging quality and improve the patients' care in imaging session.

ELIGIBILITY:
Inclusion Criteria:

* suspecting to have experienced stroke or cerebral ischemia and needed to undergo brain imaging and vascular imaging including CT or MRI
* no history of kidney failure
* a minimum age of 18 years
* obtained written informed consent

Exclusion Criteria:

* severe movement artifacts
* incidental finding of tumor lesion or craniocerebral surgery history
* poor imaging failed to perform deep learning method
* women who pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have experienced stroke or cerebral ischemia and undergone brain imaging and vascular imaging.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The performance of deep enhanced imaging in lesion detection and diagnosis | 1 year
  The performance of deep enhanced imaging in lesion detection and diagnosis, including imaging quality, accuracy, sensitivity and specificity in lesion detection and imaging diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lou Xin, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China